CLINICAL TRIAL: NCT00272610
Title: Topical Vitamin A (All-trans Retinol) Versus Vehicle Cream in the Treatment of Aged Skin
Brief Title: Topical Vitamin A Versus Vehicle Cream in the Treatment of Aged Skin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: Derm 443
Record Dates: First submitted 2006-01-03; First posted 2006-01-06 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2006-09

CONDITIONS: Skin Aging; Purpura
Keywords: Skin Aging; Bateman's Purpura
MeSH Terms: conditions — Purpura

INTERVENTIONS:
Drug: 0.4% Retinol Cream

SUMMARY:
The objectives of this study are to evaluate the safety and efficacy of 0.5% retinol (Vitamin A) versus it's vehicle cream in the treatment and prevention of skin aging and Bateman's Purpura (bruising).

DETAILED DESCRIPTION:
Human skin becomes thinner and looses its elasticity with increasing age. These features of intrinsic skin aging are due to reduction in collagen synthesis with a concomitant increase in collagen and elastic fiber breakdown by matrix metalloproteinase (MMPs). In addition to these changes that occur simply from the passage of time, skin that is chronically exposed to the sun undergoes accelerated aging process referred to as photoaging. Here sun causes further alterations in dermal matrix by transiently inducing MMPs with each irradiation. Bateman's purpura (BP) is a bruised lesion that is commonly seen on the sun-exposed extensor surfaces of forearms and hands in elderly individuals. It is of no medical significance. However, to those afflicted, BP is often a great source of distress for its unsightliness and the obvious sign of aging it represents. The pathophysiology of BP has not been rigorously studied. Its exclusive presence on the sun-exposed surfaces of frequently traumatized areas suggests that photoaging associated loss of supporting structures around cutaneous blood vessels render the vessels easily torn by shearing injuries, thus causing purpura.

Topical use of tretinoin (RA) 0.1% cream has been demonstrated to improve clinical as well as histologic changes associated with photodamaged skin. Improvement in skin wrinkles by RA appears to be related to dermal changes. RA causes accumulation of epidermal and dermal TGF-alpha 1, a cytokine known to stimulate the synthesis of collagen I and VII, both of which, by ultrastructural criteria, are increased by RA in photodamaged skin. In fact, induction of dermal collagen formation by topically applied RA has been demonstrated in animal studies, and this has been confirmed in human studies. Therefore, it is postulated that topical treatment of BP prone skin with RA would buttress up cutaneous blood vessels by increasing the supporting collagenous structures around them. Such vessels ought to withstand shearing forces better, which would lead to some protection against the development of BP.

Retinol is a precursor to RA. When applied to human skin, it mediates all the effects that RA causes, but does so with much less skin irritation. Therefore, it is expected to be better tolerated by elderly skin than RA. In a seven day treatment study of elderly patients, retinol has been shown to induce mRNA levels of procollagen molecules in human skin in vivo. Therefore, it is hypothesized to improve the thin skin of elderly by increasing the synthesis of more collagen in both the photoaged, and hence improve BP, and the intrinsically aged human skin without causing significant irritant skin reaction.

ELIGIBILITY:
Inclusion Criteria:

* Male and female
* 70 years of age or older
* history of Bateman's purpura on arms
* Relatively good general health and able to perform daily tasks

Exclusion Criteria:

* Sensitivity to any formulation ingredients
* History of Cardiovascular disease with continuing deficits (example: partial paralysis)
* Participated in any clinical trials within last 30 days
* Topical steroids or other drugs two weeks prior to study entry (short-term application of topical antimicrobials is allowed)
* Hormone replacement therapy within last 6 months.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50
Dates: Start 2000-09; Study Completion 2002-02

PRIMARY OUTCOMES:
Surface Roughness
Fine wrinkles
Hyperpigmentation
Purpura

SECONDARY OUTCOMES:
Collagen content of skin biopsies
Glycosaminoglycan expression
CRABP-II expression

CONTACTS AND LOCATIONS:
Overall Officials: John J Voorhees, MD, Study Chair — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Kafi R, Kwak HS, Schumacher WE, Cho S, Hanft VN, Hamilton TA, King AL, Neal JD, Varani J, Fisher GJ, Voorhees JJ, Kang S. Improvement of naturally aged skin with vitamin A (retinol). Arch Dermatol. 2007 May;143(5):606-12. doi: 10.1001/archderm.143.5.606. PMID 17515510